CLINICAL TRIAL: NCT04717102
Title: Evaluating the Use of Desflurane in Patients Undergoing Spinal Surgery: A Randomized Controlled Trial Using 0.5 and 0.75 MAC Desflurane
Brief Title: Evaluating the Use of 0.5 and 0.75 MAC Desflurane in Patients Undergoing Spinal Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Changi General Hospital (Other)
Responsible Party: Principal Investigator, Leong Wai May, Senior Consultant, Changi General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Desflurane01
Record Dates: First submitted 2021-01-13; First posted 2021-01-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Anesthesia
Keywords: evoked potentials; spinal surgery; desflurane
MeSH Terms: interventions — Desflurane

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 0.75 MAC desflurane (Experimental): The effects of 0.75 MAC desflurane on the amplitude and latency of evoked potentials in spinal surgeries will be examined.
  Interventions: Drug: 0.75 MAC desflurane; Drug: 1.0 MAC desflurane
- 0.5 MAC desflurane (Active Comparator): The effects of 0.5 MAC desflurane on the amplitude and latency of evoked potentials in spinal surgeries will be examined.
  Interventions: Drug: 0.5 MAC desflurane; Drug: 1.0 MAC desflurane

INTERVENTIONS:
Drug: 0.5 MAC desflurane — Following induction of anesthesia by propofol, the patients will be maintained on 0.5 MAC desflurane with remifentanil infusion during spinal surgery.
  Other Names: 0.5 MAC desflurane (Suprane)
  Arms: 0.5 MAC desflurane
Drug: 0.75 MAC desflurane — Following induction of anesthesia by propofol, the patients will be maintained on 0.75 MAC desflurane with remifentanil infusion during spinal surgery.
  Other Names: 0.75 MAC desflurane (Suprane)
  Arms: 0.75 MAC desflurane
Drug: 1.0 MAC desflurane — On completion of the neuromonitoring phase of surgery, the patients will be maintained on 1.0 MAC desflurane with remifentanil infusion.
  Other Names: 1.0 MAC desflurane (Suprane)

SUMMARY:
Background: Somatosensory- (SSEPs) and motor-evoked potentials (MEPs) are commonly used as an intraoperative neurophysiologic monitoring tool to detect aberrations to the spinal cord integrity during spinal surgery. Inhalational anaesthetic agents have a significant influence on evoked potentials by suppressing the amplitude and prolonging the latency. Evidences suggest that total intravenous anaesthesia (TIVA) is superior to inhalation anaesthesia for neuromonitoring in spinal surgery, and support the use of up to 0.5 minimum alveolar concentration (MAC) of inhalational anaesthetic agents in these procedures.

Methods: Patients undergoing spinal surgeries will be prospectively recruited and be induced with TIVA at baseline of the evoked potentials. They will be randomized to receive balance anaesthesia with A) Desflurane MAC 0.5+remifentanil, or B) Desflurane MAC 0.75+remifentanil until the end of surgery. Influence of 1.0 MAC desflurane on the evoked potentials after the completion of surgery will also be studied.

Desired Results: Endpoints include the changes to the amplitude and latency of SSEPs and MEPs with 0.5 and 0.75 MAC desflurane. The findings will indicate the safety of desflurane at the studied concentrations for spinal surgeries, and substantial savings with the use of desflurane instead of TIVA.

DETAILED DESCRIPTION:
Recording of Evoked Potentials characteristics:

The following characteristics of the evoked potential signals will be recorded:

* Amplitude: Size of the response, measured in microvolts (μV)
* Latency: Speed of the response, measured in milliseconds (ms)
* Morphology: Appearance of the response - Simple/Complex wave shape Baseline evoked potentials will be recorded at various points of surgery.

Anaesthesia variables:

At the time of recording of evoked potentials:

- Intraoperative temperature, blood pressure, ETCO2, anaesthesia depth - bispectral index monitoring (BIS), remifentanil TCI, MAC of desflurane, Train of Four, volume of propofol and remifentanil until randomization, total volume of desflurane and remifentanil used, anaesthetic medications used, FiO2, SpO2

Patient characteristics:

- Age, gender, race, weight, BMI, medications used, haematocrit, preop blood glucose (for Diabetics)

Safety considerations:

'Recommended standards for intraoperative monitoring of somatosensory evoked potentials', Guideline 11B of the American Clinical Neurophysiology Society (2009) and 'Intraoperative motor evoked potential monitoring - A position statement by the American Society of Neurophysiological Monitoring' will form the basis of the safety aspects of the study.

Conduct of Anaesthesia:

* The induction of anaesthesia will be achieved using targeted propofol and remifentanil infusions (TIVA). Muscle relaxants atracurium, rocuronium or suxamethonium will be used to facilitate intubation.
* Anaesthesia will be maintained on TIVA until the patient has recovered from muscle relaxant. Baseline characteristics (BC1) of the evoked potentials in TIVA will be obtained at this stage.
* Once the BC1 has been obtained, the patients will be randomized to two groups:

Group A- Anaesthesia maintained with 0.5 MAC desflurane/remifentanil infusion Group B- Anaesthesia maintained with 0.75MAC desflurane/remifentanil infusion

* Baseline characteristics 2 (BC2) will be obtained and the decision to proceed with 0.5 or 0.75 MAC desflurane made.
* On completion of the neuromonitoring phase of surgery, as defined by completion of instrumentation and start of closure, all patients in Group A and B will be maintained with 1.0 MAC desflurane with remifentanil infusion. Baseline characteristics 3 (BC3) will be recorded at this stage.
* The remifentanil infusion will be titrated at various stages of surgery to maintain a stable BIS and will also be based on haemodynamic variables.

All patients will get additional analgesics and antiemetics as deemed necessary. Post-operative recovery will follow the standard industry norms.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 21 years old, scheduled for spinal surgery.
* Patients who require SSEP/MEP and with no neurological deficits.
* Patients of American Society of Anesthesiologist I-III physical status.
* Consenting patients.
* Elective procedures.

Exclusion Criteria:

* Patients with sensory or motor deficits preoperatively.
* Patients with significant cardiovascular and/or respiratory disease.
* Emergency procedures.
* Cord injury secondary to trauma.
* Non-consenting patients.
* Category A patients (Prisoners).
* Patients with previous stroke.
* Patients with Hep C, HIV.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2024-03-27 (Actual); Study Completion 2024-03-27 (Actual)

PRIMARY OUTCOMES:
Effect of 0.5 MAC desflurane on evoked potentials - Amplitude (microvolts) | During surgery
  Amplitude of somatosensory- and motor- evoked potentials with use of 0.5 MAC desflurane
Effect of 0.5 MAC desflurane on evoked potentials - Latency (milliseconds) | During surgery
  Latency of somatosensory- and motor- evoked potentials with use of 0.5 MAC desflurane
Effect of 0.5 MAC desflurane on evoked potentials - Morphology (appearance of the response) | During surgery
  Morphology of somatosensory- and motor- evoked potentials with use of 0.5 MAC desflurane
Effect of 0.75 MAC desflurane on evoked potentials - Amplitude (microvolts) | During surgery
  Amplitude of somatosensory- and motor- evoked potentials with use of 0.75 MAC desflurane
Effect of 0.75 MAC desflurane on evoked potentials - Latency (milliseconds) | During surgery
  Latency of somatosensory- and motor- evoked potentials with use of 0.75 MAC desflurane
Effect of 0.75 MAC desflurane on evoked potentials - Morphology (appearance of the response) | During surgery
  Morphology of somatosensory- and motor- evoked potentials with use of 0.75 MAC desflurane

SECONDARY OUTCOMES:
Effect of 1.0 MAC desflurane on evoked potentials - Amplitude (microvolts) | intraoperative
  Amplitude of somatosensory- and motor- evoked potentials with use of 1.0 MAC desflurane
Effect of 1.0 MAC desflurane on evoked potentials - Latency (milliseconds) | intraoperative
  Latency of somatosensory- and motor- evoked potentials with use of 1.0 MAC desflurane
Effect of 1.0 MAC desflurane on evoked potentials - Morphology (appearance of the response) | intraoperative
  Morphology of somatosensory- and motor- evoked potentials with use of 1.0 MAC desflurane

CONTACTS AND LOCATIONS:
Overall Officials: Wai May Leong, MMed, Principal Investigator — Changi General Hospital
Locations (1):
- Changi General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hasan MS, Tan JK, Chan CYW, Kwan MK, Karim FSA, Goh KJ. Comparison between effect of desflurane/remifentanil and propofol/remifentanil anesthesia on somatosensory evoked potential monitoring during scoliosis surgery-A randomized controlled trial. J Orthop Surg (Hong Kong). 2018 May-Aug;26(3):2309499018789529. doi: 10.1177/2309499018789529. PMID 30058437
- [Background] Sloan TB, Toleikis JR, Toleikis SC, Koht A. Intraoperative neurophysiological monitoring during spine surgery with total intravenous anesthesia or balanced anesthesia with 3% desflurane. J Clin Monit Comput. 2015 Feb;29(1):77-85. doi: 10.1007/s10877-014-9571-9. Epub 2014 Mar 19. PMID 24643708
- [Background] Macdonald DB, Skinner S, Shils J, Yingling C; American Society of Neurophysiological Monitoring. Intraoperative motor evoked potential monitoring - a position statement by the American Society of Neurophysiological Monitoring. Clin Neurophysiol. 2013 Dec;124(12):2291-316. doi: 10.1016/j.clinph.2013.07.025. Epub 2013 Sep 18. PMID 24055297